CLINICAL TRIAL: NCT05219708
Title: Impact of a High Energy and High Protein Nutrition Supplementation Intervention on Outcomes in Patients With Advanced Heart Failure
Brief Title: High Calorie High Protein Nutrition Supplementation in Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mathew S. Maurer, MD, Professor of Cardiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAT7938
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calorie and protein nutritional supplementation (Experimental): Study participants randomized to the intervention will receive 30 days worth of the nutritional supplement (i.e. Ensure Original) to be consumed twice per day in between meals in addition to standard of care for heart failure.
  Interventions: Dietary Supplement: Calorie protein supplement
- Control (Active Comparator): The control group will receive standard of care for heart failure.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Calorie protein supplement — Participants assigned to the intervention group will receive the calorie and protein supplement (i.e. Ensure Original) to be consumed twice daily between meals for 30 days in addition to standard of care for heart failure
  Arms: Calorie and protein nutritional supplementation
Other: Control — Standard of care for heart failure
  Arms: Control

SUMMARY:
In this study, the investigators will determine the impact of a high calorie and high protein nutrition supplementation strategy on quality of life in participants with advanced heart failure. The investigators hypothesize that participants with advanced heart failure who receive the high calorie high protein nutrition supplementation strategy will experience an improvement in quality of life compared to those patients that receive usual care.

DETAILED DESCRIPTION:
This is a single center, prospective randomized open with blinded endpoint (PROBE) trial with an individual follow-up time of 30 days duration designed to determine the impact of a high calorie high protein nutritional supplementation strategy on quality of life and functional outcomes in adults with malnutrition advanced systolic heart failure. 48 participants will be randomized in a stratified fashion by gender and Subjective Global Assessment (SGA) class (B versus C). Study subjects will receive a calorie and protein nutritional supplement, Ensure Original, manufactured by Abbott laboratories for 30 days after hospital discharge. The study site will be Columbia University Irving Medical Center. Investigators will be blinded to group assignment and dietary recalls until the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Hospitalized at Columbia University Irving Medical Center/New York Presbyterian Hospital
* Left ventricular ejection fraction <=40%
* At least mild malnutrition as determined by the Subjective Global Assessment (SGA)

Exclusion Criteria:

* Inability to eat orally
* Inability to eat independently
* History of dysphagia
* Allergy to nutritional supplement
* Need for inotrope and/or mechanical support at hospital discharge
* Listed for heart transplant
* Insulin dependent diabetes and/or most recent A1c >7%
* Having two or more results of a serum potassium >5.0 mmol/L during hospitalization or history of serum potassium >6.0 mmol/L, and/or at an excessive risk of hyperkalemia as judged by the investigators
* Severe renal insufficiency (estimated glomerular filtration rate <30 ml/min/1.73m^2 at discharge)
* Cirrhosis
* History of bariatric surgery
* Nursing home residence
* History of persistent noncompliance with treatment recommendations as judged by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Score | Up to 30 days
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a self-administered questionnaire to assess quality of life in heart failure. Scores range from 0-100 with a higher score indicating better quality of life.

OTHER OUTCOMES:
Change in handgrip strength | Up to 30 days
  Handgrip strength as measured by Jamar Hydraulic Hand Dynamometer
Change in Short Physical Performance Battery (SPPB) Score | Up to 30 days
  SPPB measures functional capacity. Scores range from 0 (lowest physical performance) to 12 (highest physical performance).

CONTACTS AND LOCATIONS:
Overall Officials: Mathew S. Maurer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No